CLINICAL TRIAL: NCT06715033
Title: Relationship Between Ankle Planterflexors Peak Torque and Balance in Patients With Functional Ankle Instability
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Mohammed Mahmoud Khafaga, Demonstrator at AHUC, Cairo University
Other Study IDs: P.TREC/012/005361
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Functional Ankle Instability
Keywords: Calf Muscles; Isokinetic; Y balance; Side hop

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Group A (Experimental): 34 affected ankles of both genders diagnosed with functional ankle instability (FAI) who met the inclusion criteria. Their ages ranged from 18 to 25 years, and the patients had a history of initial injury, ongoing bouts of instability, and ratings of patient-perceived function and disability.
  Interventions: Diagnostic Test: y balance and SLS
- 2: Group B (Control): This group consisted of 34 matched non-affected ankles in the study.
  Interventions: Diagnostic Test: y balance and SLS

INTERVENTIONS:
Diagnostic Test: y balance and SLS — for assessment of static and dynamic balance
  Other Names: side hop

SUMMARY:
This study attempted to:

1. Investigate the difference in calf muscle strength (concentric and eccentric) between affected limb with instability and non-affected limb.
2. Assess the relationship between the severity of ankle instability and calf muscle strength (concentric and eccentric) at velocity (60 and 120◦/s) in patients with functional ankle instability?
3. Investigate the relationship between calf muscle strength (concentric and eccentric) deficit and functional performance in functional ankle instability.

DETAILED DESCRIPTION:
Statement of the problem Was there a difference in calf muscle strength (concentric and eccentric) between the affected limb with instability and the non-affected limb? Was there a relationship between the severity of ankle instability and calf muscle strength (concentric and eccentric) at velocities of 60 and 120°/s in patients with functional ankle instability? Was there a relationship between calf muscle strength (concentric and eccentric) deficits and functional performance in patients with functional ankle instability?

Purpose of The Study

This study attempted to:

1. Investigate the difference in calf muscle strength (concentric and eccentric) between affected limb with instability and non-affected limb.
2. Assess the relationship between the severity of ankle instability and calf muscle strength (concentric and eccentric) at velocity (60 and 120◦/s) in patients with functional ankle instability?
3. Investigate the relationship between calf muscle strength (concentric and eccentric) deficit and functional performance in functional ankle instability.

Significance of study Chronic ankle instability is recognized as one of the most common lower-extremity disorders encountered by orthopedic physical therapists The prevalence of CAI varies from 0.7% to 1.1% in young people, 20% in student-athletes, 23.4% in collegiate and high school athletes, and 29% in high school pupils Incidents of CAI are roughly 7/1000 person-years in the general population and up to 45/1000 person-years in those who engage in physical activity Chronic ankle instability may develop as a result of improper post-injury management and a lack of medical attention.

There is an urgent need for diagnostic and measurement methods to pinpoint and follow people who are at risk of CAI.

Lack of research on plantar flexors and additional studies evaluating isokinetic ankle torque values are necessary.

Different studies examined ankle muscles (evertors, invertors, dorsiflexors, and plantar flexors) eccentric contractions only, and no one study examined calf muscle concentric and eccentric contractions in CAI.

Several studies have provided evidence that concentric plantarflexor strength are impaired CAI.

Insufficient strength of plantarflexor may alter performance, hence this study will instruct strength of calf muscles to prevent ankle injury.

Effective evaluation is the first step toward effective treatment; earlier research limited the fundamental basis for rehabilitation after ankle injury by failing to identify variables linked to symptoms of ankle instability.

Functional tests are useful as a guide for rehabilitation outcomes because they can identify deficiencies in muscular strength and functional performance limits. So far, there is no gold standard for the assessment and treatment of chronic ankle instability.

Up to the authors' knowledge, there is limited evidence about calf muscle strength, which is neglected in rehabilitating chronic ankle instability. Therefore, this study will assess calf muscle strength in patients with functional ankle instability. This trial will guide physical therapists to address calf muscle strength in assessment and treatment procedures for managing FAI.

Hypotheses of the Study

1. There was no statistical relationship between the severity of functional ankle instability and calf muscle strength (concentric and eccentric) in patients with ankle instability.
2. There was no statistically significant difference in calf muscle strength (concentric and eccentric) at velocities of 60°/s and 120°/s between the affected limb with ankle instability and the non-affected limb.
3. There was no statistical relationship between calf muscle strength (concentric and eccentric) and dynamic balance in patients with ankle instability.
4. There was no statistical relationship between calf muscle strength (concentric and eccentric) and static balance in patients with ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

Subjects' selection was based on the following criteria:

1. Age ranged from 18 to 25 years
2. The body mass index was 18.5 to 24.9 kg/m2
3. History of at least one unilateral lateral ankle sprain that needed to be immobilized for three days or longer
4. At least one recurring sprain in the three to six months before study participation.
5. FAI if their total score is 11 or above by IdFAI.

Exclusion Criteria:

* Exclusion criteria

Subjects were excluded if they had any of the following criteria:

1. Previous Ankle surgery.
2. Patients with bilateral ankle instability.
3. Syndesmotic and medial ankle sprain .
4. Severe ankle arthritis.
5. Neurological disorders affect ankle function.
6. No history of ankle fractures .

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: age sex
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Arabic version of the Identification of Functional Ankle Instability questionnaire (IdFAI-AR) | 1 session
  asses of FAI

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Khafaga, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Abdelkader NA, Khafagaa MM, Aziz MZ. The gastrocnemius and soleus muscles deficits in functional ankle instability: an observational study. BMC Musculoskelet Disord. 2025 Nov 14;26(1):1046. doi: 10.1186/s12891-025-09286-4. PMID 41239273